CLINICAL TRIAL: NCT00519272
Title: A Prospective Study Examining the Barriers to Care for Harris County Cervical Cancer Patients
Status: Terminated | Type: Observational
Why Stopped: Requested by PI during yearly Continuing Review
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0530
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Cervix; Precancerous Lesions; Cervical carcinoma in situ; CIS; Early cervical cancer detection and treatment; Barriers to Care; Harris County; Questionnaire
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical Cancer Care Questionnaires: New cervical cancer patients through stage IVB presenting to the LBJ Gyn-Onc Clinic.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Series of surveys to be completed at the time of diagnosis and within one month after completion of treatment, taking approximately 45 minutes each time.
  Other Names: Survey

SUMMARY:
The goal of this behavioral research study is to look at the reasons that may prevent women from getting early treatment for their cervical cancer.

DETAILED DESCRIPTION:
Little is known about what prevents women with cervical cancer from getting early and possibly curative treatment. This study consists of a series of questionnaires that ask questions about religion; coping; access to health care; physical, emotional, and spiritual well-being; understanding of health questions; control; fear; anxiety; and other health beliefs to determine why some women delay coming in for check-ups and why some women do not complete their treatments. It is thought that health beliefs influence behavior practices and that by identifying these issues, things can be done to improve the health condition and results for these patients.

You will be asked to complete a series of questionnaires at 2 specific time points: The first time point will be before treatment begins and the second time point will be within a month following completion of treatment.

Filling out the questionnaires should take about 45 minutes each time. You should have adequate time to complete these questionnaires during your clinic appointment.

If you want to take part but are too ill to complete the questionnaires, you will be provided a pre-addressed, stamped envelope, so that you can mail them back to the study staff at your earliest convenience.

This is an investigational study. This is an investigational study. Up to 150 patients will be enrolled at Lyndon B. Johnson General Hospital.

ELIGIBILITY:
Inclusion Criteria:

1) All newly diagnosed cervical cancer patients through Stage IVB presenting to the Lyndon B. Johnson General Hospital (LBJ) Gynecologic Oncology Clinic.

Exclusion Criteria:

1) Patients who are not English or Spanish speaking.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed cervical cancer or precancerous lesions (CIS) seen in the Gynecologic-Oncology or Colposcopy Clinic at Lyndon B. Johnson General Hospital in Houston, Texas.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-07-21 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Issues preventing access to early cervical cancer detection and treatment among Harris County cervical cancer patients. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Lois M. Ramondetta, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Lyndon B. Johnson General Hospital, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org